CLINICAL TRIAL: NCT02400554
Title: Yappalli - The Road to Choctaw Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Karina Walters, Associate Dean for Research; William P. and Ruth Gerberding Endowed University Professor, University of Washington
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: STUDY00001641; R01DA037176 (NIH)
Record Dates: First submitted 2015-03-17; First posted 2015-03-27 (Estimated); Last update posted 2022-11-03 (Actual); Status verified 2021-09

CONDITIONS: Obesity; Substance Abuse
Keywords: Indian, North American; Oklahoma; Female; health promotion
MeSH Terms: conditions — Obesity; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Wait List Control (No Intervention): Participants wait one year before receiving the intervention. Three assessments are taken over this period: Month 3, Month 9, and Month 12.
- Yappalli (Experimental): Yappalli: Participants attend a 12-month behavioral intervention.
  Interventions: Behavioral: Yappalli

INTERVENTIONS:
Behavioral: Yappalli — Month 1-3: Up to 8 group sessions on Choctaw history, traditions, cultural systems, & women's roles. Up to 3 individual Motivational Interviewing (MI) sessions to identify community leadership & personal change goals on the main outcome.
  Month 2: Overnight Culture Camp to strengthen group cohesion & synthesize goals.
  Month 3: Walk for a week on the Choctaw Trail of Tears, upon completion make a commitment to conduct a community-wide event based on personal & leadership goals & experience on the Trail.
  Months 3-12: Up to 6 group meetings to plan community leadership events related to ATOD & obesity prevention. Includes: digital storytelling training to create a story related to ATOD & obesity prevention & an individual MI booster session to revise their personal & community leadership goals.
  Month 12: Share digital stories & community event experiences & undergo a ceremony to transition to health leaders within their communities.
  Arms: Yappalli

SUMMARY:
This is an obesity and alcohol, tobacco, and other drug (ATOD) use risk prevention and health leadership program. This project will include 150 at-risk adult Native women across 5 communities (30 women from each community) in the Choctaw Nation of Oklahoma. The intervention targets individual behavioral change relative to ATOD and obesity prevention and simultaneously provides behavioral skills for health promotion leadership.

Investigators will conduct a longitudinal study using a cluster randomized stepped-wedge design to evaluate the intervention impact on ATOD and obesity prevention primary aims of: (1) substance use harm reduction and ATOD use and intentions to use; and (2) reduction in weight/body mass index (BMI) and increase in leisure-time physical activity/physical activity (LTPA/PA) and healthful food habits. Specifically, investigators will ask participants to participate in up to eight group sessions (based on a curriculum drawing on cultural teachings around health and behavioral change); attend up to three Motivational Interviewing individual sessions (to identify individual behavioral change goals); attend a two-day overnight culture and Trail prep camp; participate in camping and walking for up to 10 days on the Trail; and attend up to six post-walk meetings (to develop community health events). All five communities will also be asked to complete a baseline health assessment as well as three follow up assessments over the course of the year. Additionally, communities 2-5 will participate in three pre-intervention health assessments. This intervention integrates components of motivational interviewing, information-motivation-behavior, and a leadership development framework for adults. It targets individual behavioral change relative to ATOD and obesity prevention and simultaneously provides behavioral skills for health promotion leadership within their respective communities.The project addresses a critical public health issue among a group experiencing considerable health disparities and strengthens the research infrastructure in partnership with the Tribe. If efficacious, it has the potential for widespread dissemination and could be generalizable to other chronic co-occurring mental health and physical health conditions.

DETAILED DESCRIPTION:
Study Design:

Investigators will conduct a 5-community longitudinal study using a cluster randomized stepped-wedge design to evaluate the intervention impact on alcohol, tobacco, and other drug (ATOD) and obesity prevention primary aims of: (1) substance use harm reduction, overall ATOD use and intentions to use; and (2) weight/body mass index (BMI) change as well as the effect on leisure-time physical activity/physical activity (LTPA/PA), and healthful food habits among adult Choctaw women at risk for obesity and ATOD. The cluster randomized stepped-wedge design is a type of cross-over study in which clusters of women from each community cross over to the intervention arm at randomly assigned time points (one time per year, per community).

Sequence and Timing of Study Procedures:

Randomization: Investigators have created five regional communities and within each community a convenience sample will be drawn. Each site has been randomly assigned to start the intervention at a given year. Randomization occurs only to determine the year each community enters the study. Community 1 will begin the intervention immediately; communities 2-5 will complete three health assessments prior to beginning the intervention. These will occur at the same time of post-walk assessments for the community currently in the intervention (i.e. community 2 does health assessments in the same months community 1 does post-walk assessments and then begins the intervention in Year 2.)

Recruitment and Screening of Participants:

Recruitment strategies:

* Referrals from staff from Choctaw Nation of Oklahoma (CNO) project staff, staff at Choctaw Nation Health Services Authority (CNHSA), Community Advisory Council members, health providers, and general community members. They will provide potential participants with a flyer and encourage women to call if interested.
* The following strategies will be used as necessary: posting flyers in community health clinics, stores, community centers, and other locations identified by our community advisors; and posting flyers in the tribal newspaper, other local news outlets, and on a study Facebook page.
* Recruitment materials will invite American Indian/Alaska Native women who are interested in participating in the research study to call a dedicated, toll-free phone number or the project number at Choctaw Nation.

Screening:

* Participants can opt for a phone or in-person screen using the same script.
* CNO study staff will answer and return phone calls and conduct the screens. Indigenous Wellness Research Institute (IWRI) staff will conduct eligibility screens on the phone as needed.
* Women screened out will be given a community resource list. Phone screeners will offer to mail or email the list.
* If a person is eligible, but declines to participate, they will be given a brief one-item exit question regarding general reason for non-participation.
* Eligible women who agree to participate will be asked to schedule their baseline assessment.

Participants will receive reminders by email, text or phone 2 days before, the day before, and the day of any meetings, assessments, or events.

Consent and Baseline Assessment:

The baseline assessment consists of a brief physical health assessment and a computer-assisted behavioral health survey administered by study staff. The physical health assessment is a non-invasive procedure that involves the measurement of BMI (with portable digital weight scale and height measure) and blood pressure. The computer-assisted behavioral health survey will ask a series of questions and take under 90 minutes to complete.

After consent is obtained, CNO study staff will set up the study laptop and headphones that the participant will use to enter their responses to the questionnaire. The variable matrix includes instructions, prompts, response scales, and references for all measures used for each behavioral health assessment.

Group Sessions/Yappalli Curriculum (Months 1-3) Participants will attend up to eight group sessions. The curriculum for these sessions includes: learning about Choctaw history, traditions,and cultural systems as well as women's roles (e.g., Treaty of Dancing Rabbit Creek); participating in cultural activities (e.g., stickball or social dances); developing traditionally-based materials (e.g., walking sticks); and using cultural metaphors for behavioral changes (e.g., 4 pillars of wellness-mind, body, spirit, emotion)). Experiential, outdoor activities are incorporated to promote group cohesion, improve relational worldviews, and connectedness to nature and the environment. Examples include activities on an outdoor ropes course maintained and managed by CNHSA or increasing LTPA/PA by walking or gardening.

Motivational Interviewing Individual Sessions (Months 1-3) In up to three sessions, participants will identify personal change goals on the main outcome variables as well as community leadership goals. These sessions will target four areas: increasing physical activity or movement; reducing or eliminating "junk" snack foods, sweets, and sugared soft drinks; decreasing addiction and or potential to misuse tobacco, alcohol or other substances and food; and increasing community leadership skills.

Culture Camp (Month 2) In this two-day, overnight camp participants will practice camping and being outdoors (e.g., setting up tents, trying out new shoes and equipment, etc.) and begin to strengthen group cohesion prior to embarking on the Trail. It is also designed to synthesize goals and cultural values discussed in the group and individual sessions.

Trail of Tears Walk (Month 3) Participants will gather at a location in Oklahoma before driving to a starting point at the Mississippi/Arkansas border then follow one of the routes of the Choctaw Trail of Tears through Arkansas and back into Oklahoma. They will walk on average 8-10 miles per day and travel by van for a portion of the trail to a different campsite each day. At the end of the trip, the walkers will have walked approximately 60-80 miles over the 260 mile route. On the last night of the Trail, participants will make a vow to conduct a community-wide event (based on personal and leadership goals and experience on the Trail) within nine months. Note: a support van will travel along with walkers so that they could walk as many minutes or miles they feel comfortable doing (e.g., from 10 mins. Less than a quarter mile to 10 miles).

Post-Walk assessments (Months 3-12) Three follow-up health assessments will occur: one immediately post-walk in Month 3, one in Month 9, and one in Month 12. These behavioral health assessments will be collected in the same manner and include a similar set of measures as the baseline assessment. The physical health assessments will also be conducted in the same manner as the baseline assessment.

Post-Walk Group Meetings (Months 3-12) Participants will attend up to six group meetings to plan community leadership events (investigators provide a small budget for the women to create a community event such as a community food garden). Specific meetings include: at three months post-walk a digital storytelling training to create a story related to ATOD and obesity prevention and their personal experiences; and at six months post-walk an individual MI booster session to revise their personal vows/goals and community leadership goals.

Final Community Event (Month 12) Participants will share digital stories and/or community event experiences and undergo a naming ceremony as they transition to health leaders within their communities. They will be given the option to become a member of one of seven Choctaw health promotion societies on which the intervention is based to continue their health promotion leadership efforts after their participation in the project ends.

ELIGIBILITY:
Inclusion Criteria:

* Self-identify as women
* Be enrolled in the Choctaw Nation of Oklahoma
* Reside in the designated county
* Be 18 years of age or older
* Have tried any tobacco, alcohol, or drugs OR ever felt out of control with any food in past 5 years
* Be able to walk unassisted for at least 10 minutes

Exclusion Criteria:

* Women who are actively using opioids (i.e., heroin) methamphetamines and/or abusing prescription drugs not prescribed to them (e.g., Dilaudid, Oxycontin) or alcohol dependent (5+ bottles/glasses of alcohol a day).
* Women who exhibit serious psychiatric symptoms determined by CNO trained staff.
* Women who have been suicidal in past 3 months, are currently pregnant, or are denied medical approval.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Change in Food Habits as assessed by the Yale Food Addiction Scale | Post-Walk (month 3) and Post Intervention (month 12)
  Yale Food Addiction Scale - continuous measure items
Weight Change | Post-Walk (month 3) and Post Intervention (month 12)
  Investigators will assess weight change for each individual
Changes in Physical Activity assessed using items from the California Health Interview Survey | Post-Walk (month 3) and Post Intervention (month 12)
  Investigators will assess changes in physical activity and leisure time activity in participants using items from the California Health Interview Survey
Change in Alcohol Use as assessed by the Alcohol Use Disorders Identification Test. | Post-Walk (month 3) and Post Intervention (month 12)
  Assess changes in alcohol use (frequency, amount, consequences and context) using the Alcohol Use Disorders Identification Test.
Change in Other Substance Use as assessed by the Phen-X toolkit | Post-Walk (month 3) and Post Intervention (month 12)
  Phen-X toolkit for 30-Day Use (for items that are applicable)

CONTACTS AND LOCATIONS:
Overall Officials: Karina L Walters, PhD, Principal Investigator — University of Washington; Kristie Brooks, Principal Investigator — Choctaw Nation of Oklahoma; Michelle Johnson-Jennings, PhD, Principal Investigator — University of Washington
Locations (1):
- Choctaw Nation of Oklahoma, McAlester, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No